CLINICAL TRIAL: NCT07397104
Title: Validity of a Self-Reported Questionnaire for Periodontal Status in a Saudi Population: A Cross-Sectional Clinical Validation Study
Brief Title: Validity of a Self-reported Questionnaire for Periodontal Status in a Saudi Population
Status: Not yet recruiting | Type: Observational
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Abdulrahman Ahmed M. Alshehri, Principal Investigator, Universiti Sains Malaysia
Other Study IDs: F3-12-2025
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Periodontal Diseases; Periodontitis; Gingivitis
Keywords: Periodontal disease; Validity; self-reported
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingivitis | interventions — Reference Standards

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults attending screening appointments (self-report + same-visit clinical exam): Participants scheduled for screening appointments at Asir Specialized Dental Center will complete a self-reported periodontal questionnaire (CDC-AAP items). During the same visit, a trained clinician will perform a standardized clinical periodontal examination to determine periodontal status (full mouth periodontal examination based on CDC/AAP and EFP case definitions). Questionnaire results will be compared with the clinical findings to evaluate validity.
  Interventions: Other: Self-reported periodontal questionnaire and clinical periodontal examination (reference standard)

INTERVENTIONS:
Other: Self-reported periodontal questionnaire and clinical periodontal examination (reference standard) — Data collection procedures to validate questionnaire-based periodontal status; no therapeutic intervention is assigned.

SUMMARY:
This observational study will evaluate the accuracy of a self-reported periodontal questionnaire in adults attending screening appointments in Abha, Saudi Arabia. Participants will complete the questionnaire and then undergo a same-visit clinical periodontal examination. The study will compare questionnaire-based results with clinical examination findings to assess diagnostic accuracy and agreement.

DETAILED DESCRIPTION:
This observational, cross-sectional clinical validation study will assess the validity of a self-reported periodontal questionnaire (CDC-AAP self-report items) among adults attending scheduled screening appointments at Asir Specialized Dental Center in Abha, Saudi Arabia. At the screening visit, participants will complete the self-reported questionnaire. During the same visit, trained clinicians will perform a standardized full mouth clinical periodontal examination, which will serve as the reference standard for determining periodontal status and/or periodontal disease categories according to predefined clinical criteria in the study protocol.

The primary objective is to determine how accurately the self-reported questionnaire identifies clinically determined periodontal status. Questionnaire responses and any questionnaire-derived classification will be compared with clinical examination results to estimate diagnostic accuracy (e.g., sensitivity, specificity, and overall accuracy) and to assess agreement between questionnaire-based and clinically based classifications. Additional outcomes may include feasibility measures such as questionnaire completion rates and missing data patterns. Data will be recorded using study identifiers and stored in secure, access-controlled systems to protect confidentiality. Participation does not involve assignment to any treatment; it consists only of completing a questionnaire and undergoing a same-visit periodontal examination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to provide informed consent
* Able to complete the self-reported periodontal questionnaire
* Willing to undergo a same-visit clinical periodontal examination

Exclusion Criteria:

* Less than ten teeth present
* Any condition that makes periodontal probing unsafe, as judged by the clinician according to local policy
* Unable to complete study procedures or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from adults scheduled for dental screening appointments at Asir Specialized Dental Center, Abha, Saudi Arabia. Recruitment and all study procedures will take place at the center during the scheduled screening visit.
Sampling Method: Probability Sample
Enrollment: 291 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the self-reported periodontal questionnaire for clinically determined periodontal status | Same-visit (baseline)
  Accuracy of the self-reported periodontal questionnaire in identifying clinically determined periodontal status based on the same-visit clinical periodontal examination (reference standard). Diagnostic performance will be summarized using standard measures such as sensitivity, specificity, and area under the ROC curve, as applicable to the questionnaire-derived classification.

IPD SHARING:
Plan to Share IPD: Yes
De-identified, controlled access.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified IPD and supporting documents will be available beginning 12 months after publication of the primary results (or 12 months after study completion if not published) and will remain available for 5 years thereafter.
Access Criteria: Access will be provided to qualified researchers who submit a methodologically sound proposal (protocol/analysis plan) and obtain any required ethics approval/exemption. Approved requestors will receive de-identified participant-level data (questionnaire responses and clinical periodontal status) and selected supporting documents under a data use agreement, shared via secure transfer. No direct identifiers will be shared.